CLINICAL TRIAL: NCT05921032
Title: Low Back Pain Among Nurses: Comparison of Biomechanics, Function and Pain Across Subtypes and Effects of Exercise Intervention.
Brief Title: Comparison of Biomechanics, Function and Pain and Effects of Exercise Intervention Among Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Shazlin Shaharudin, Principal Iinvestigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: USM/JEPeM/19100637
Record Dates: First submitted 2023-04-03; First posted 2023-06-27 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2023-08

CONDITIONS: Nurses
Keywords: Kinematics; Kinetics; Human health; Spine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lumbar stabilisation exercise (LSE) (Other): Lumbar stabilisation exercise (LSE) group will perform eight weeks exercise intervention for two sessions in a week. Each session took about 45 minutes to complete. The total exercise sessions were 16 sessions. LSE group will be focused on strengthening the deep trunk stabilising muscles (i.e., transverse abdominal, internal oblique and lumbar multifidus) and control pelvis muscles.
  Interventions: Other: Exercise intervention
- Lumbar muscle strengthening exercise (LMSE) (Other): Lumbar muscle strengthening exercise (LMSE) group will perform eight weeks exercise intervention for two sessions in a week. Each session took about 45 minutes to complete. The total exercise sessions were 16 sessions. LMSE group aims to strengthen the trunk flexor and extensor muscles.
  Interventions: Other: Exercise intervention
- Control group (No Intervention): The control group will be given a diary to record their daily activities which consist of their 24 hours diet recall for 8 weeks and involvement of any physical activity throughout the 8 weeks. This diary will be collected during follow up (1 month after post-intervention). Upon completion of the trial, participants in the control group will receive either LSE or LMSE or combination of both exercises depending on their preference.

INTERVENTIONS:
Other: Exercise intervention — 8 weeks of exercise with two session in a week
  Arms: Lumbar muscle strengthening exercise (LMSE); Lumbar stabilisation exercise (LSE)

SUMMARY:
The goal of this study is to compare the effects of exercise interventions (lumbar stabilisation exercise (LSE) versus lumbar muscles strengthening exercises (LMSE)) on full body mechanics, functional disability outcomes and pain score among female nurses with chronic non-specific low back pain (CNLBP). The main questions are:

* What are the differences in full body mechanics, functional disability outcomes and pain score among female nurses with CNLBP?
* How exercise intervention affects full body mechanics, functional disability outcomes and pain score among female nurses with CNLBP?

Participants will be divided into three groups (lumbar stabilisation exercise (LSE), lumbar muscles strengthening exercises (LMSE) and control group). Exercise intervention group will be asked to perform 8 weeks of exercise intervention with :

* 3D kinematics and trunk spinal loads test
* Trunk muscle power (extensor) test
* Sit-and-reach test
* Functional disability (Roland-Morris Low Back Pain and Disability Questionnaire, RMQ)
* Pain intensity (Visual analogue scale, VAS)
* Endurance of trunk muscle test

Meanwhile control group will be given a diary to record their daily activities which consist of their 24 hours diet recall for 8 weeks and involvement of any physical activity throughout the 8 weeks.

Researchers will compare between two exercise groups to see if there is any differences in full body mechanics, functional disability outcomes and pain score across different among female nurses with CNLBP.

DETAILED DESCRIPTION:
* All participants are female nurses with age range between 20 - 55 years old from Hospital USM and have chronic LBP persisting for longer than three months.
* Randomisation of participants' selection will be conducted using computer. The allocation numbers will be generated by the computer via excel formulas to get evenly distributed names into three groups.
* The sample size is calculated using GPower software (v.3.1.9.7, Universität Düsseldorf, German) of Repeated Measure ANOVA with p value set at 0.05 and effect size is 0.75. Based on effect size, it showed that 15 participants per group are sufficient to yield 0.8 power of the study with four times of assessments (i.e., pre-intervention assessment, mid- intervention assessment, post- intervention assessment, and 1 month after intervention). By inclusion of 20% drop out rate a total of 54 participants were recruited with 18 participants per group (n=18).
* Participants need to attend at least 75% of the training session and their data will not be evaluated if they do not meet this minimum adherence level.
* All statistical analyses will be performed using Statistical Package for Social Science (SPSS) version 26.0 (IBM Inc., Armonk, New York, United States). The level of significance was set at p<0.05.All data will be tested for normal distribution via the Shapiro Wilk test. Repeated Measure ANOVA will be conducted to compare the lower extremity and trunk kinematics, endurance of trunk flexor and extensor muscles, functional disability, pain intensity values and anthropometric data across two groups at pre, middle, post and one month follow up after exercises intervention.
* All 3D kinematics and trunk spinal loads test, trunk muscle power (extensor) test, sit-and-reach test, functional disability (Roland-Morris Low Back Pain and Disability Questionnaire, RMQ), pain intensity (Visual analogue scale, VAS) and endurance of trunk muscle test will be assessed during pre assessment, middle assessment (during fourth week of exercise intervention), post assessment and after one month follow up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Female nurses from Hospital USM
* Had chronic non specific LBP persisting for longer than three months.
* Treated as outpatients of HUSM

Exclusion Criteria:

* history of cerebrovascular disease
* chronic diseases that cause long-term immobilisation
* history of previous spine surgery
* diagnosed with spinal cord disease
* history of rheumatic disease
* diagnosed with cancer
* history of neurological deficits
* history of infectious and systemic disease
* history of radicular pain due to nerve root involvement
* history of structural lesion such as spondylosis
* spondylolisthesis
* scoliosis
* kyphosis
* vertebral bone fracture

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in lumbar angle from baseline to post-intervention | through study completion, an average of 4 months
  Biomechanical data measured during walking, sit-to-stand and carrying and transferring a standard load
Change in pelvic tilt angle from baseline to post-intervention | through study completion, an average of 4 months
  Biomechanical data measured during walking, sit-to-stand and carrying and transferring a standard load
Change in hip angle from baseline to post-intervention | through study completion, an average of 4 months
  Biomechanical data measured during walking, sit-to-stand and carrying and transferring a standard load
Change in knee angle from baseline to post-intervention | through study completion, an average of 4 months
  Biomechanical data measured during walking, sit-to-stand and carrying and transferring a standard load
Change in ankle angle from baseline to post-intervention | through study completion, an average of 4 months
  Biomechanical data measured during walking, sit-to-stand and carrying and transferring a standard load
Change in back extensor muscle power from baseline to post-intervention | through study completion, an average of 4 months
  Grading of muscle strength (Oxford Scale) will be used to assess back extensor muscle power. 0/5 = no muscle movement, 1/5 = muscle movement without joint motion, 2/5 = movement with gravity eliminated, 3/5 = movement against gravity but not against resistance, 4/5 = movement against gravity and light resistance and 5/5 represents normal strength
Change in functional disability from baseline to post-intervention | through study completion, an average of 4 months
  Functional disability will be assessed by using the Roland-Morris Low Back Pain and Disability Questionnaire. Greater levels of disability are reflected by higher numbers of 24-point scale which represented 24 questions. Through analysis of serial questionnaire scores, a clinical improvement over time can be graded. For example, at the beginning of test, a participant's score was 10, and after test, her score was 2 (8 points of improvement). Therefore, the improvement percentage was 80% (8/10 x 100).
Change in pain intensity from baseline to post-intervention | through study completion, an average of 4 months
  Visual analogue scale (VAS) will be used to assess the pain intensity. The minimum values "0" referring to no pain and maximum values "10" referring to worst imaginable pain.
Change in endurance of trunk muscles from baseline to post-intervention | through study completion, an average of 4 months
  Trunk flexor muscle and extensor muscle will be tested according to the duration of the muscles contraction. Long time duration (more than 4 minutes) means the participant has no back pain.
Change in hamstrings flexibility from baseline to post-intervention | through study completion, an average of 4 months
  Flexibility of the lower back and hamstrings will be assessed by using sit and reach test. The scale will be referring to The American College of Sports Medicine (ACSM) which range from excellent to poor (in cm) according to their age.
Change in full body gravitational reaction force from baseline to post-intervention | through study completion, an average of 4 months
  Biomechanical data measured during walking, sit-to-stand and carrying and transferring a standard load
Change in full body moment from baseline to post-intervention | through study completion, an average of 4 months
  Biomechanical data measured during walking, sit-to-stand and carrying and transferring a standard load
Change in full body center of pressure from baseline to post-intervention | through study completion, an average of 4 months
  Biomechanical data measured during walking, sit-to-stand and carrying and transferring a standard load

CONTACTS AND LOCATIONS:
Overall Officials: Shazlin Shaharudin, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia Kampus Kesihatan, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moon HJ, Choi KH, Kim DH, Kim HJ, Cho YK, Lee KH, Kim JH, Choi YJ. Effect of lumbar stabilization and dynamic lumbar strengthening exercises in patients with chronic low back pain. Ann Rehabil Med. 2013 Feb;37(1):110-7. doi: 10.5535/arm.2013.37.1.110. Epub 2013 Feb 28. PMID 23525973
- [Background] Sipaviciene S, Kliziene I. Effect of different exercise programs on non-specific chronic low back pain and disability in people who perform sedentary work. Clin Biomech (Bristol). 2020 Mar;73:17-27. doi: 10.1016/j.clinbiomech.2019.12.028. Epub 2020 Jan 3. PMID 31923778